CLINICAL TRIAL: NCT00865475
Title: A Randomized Comparative Clinical Trial of ZDV + 3TC + ABC (Trizivir) vs Monotherapy With Lopinavir/R (Kaletra) in Patients With Viral Suppression on Previous Treatment With ZDV + 3TC + ABC (Trizivir) for Preventing Lipoatrophy
Brief Title: Prevention of Lipoatrophy in Patients Treated With Lopinavir/Ritonavir in Monotherapy Versus ZDV + 3TC + ABC
Acronym: KALIPO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GESIDA 6108; 2008-003438-12 (EudraCT Number); 6108 (Other: GESIDA)
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infection; HIV Infections
Keywords: HIV infection; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine, and zidovudine drug combination; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TZV (Trizivir) (No Intervention): Keeping on TZV in patients with viral suppression
- 2 (Experimental): Switching to LPV/r monotherapy
  Interventions: Drug: AZT+3TC+ABV (Trizivir); Drug: Switching to LPV/r monotherapy (Kaletra)

INTERVENTIONS:
Drug: AZT+3TC+ABV (Trizivir) — Patients on treatment with TZV and viral suppression will be randomized to keep on TZV vs switching to LPV/r monotherapy
  Other Names: LPV/r (Kaletra)
  Arms: 2
Drug: Switching to LPV/r monotherapy (Kaletra) — Patients on AZT+3TC+ABV with viral suppression will be randomized to keep on vs switching to LPV/r
  Other Names: Kaletra
  Arms: 2

SUMMARY:
The aim of this study is to measure the prevention of lipoatrophy in patients treated with Lopinavir/R in monotherapy versus ZDV + 3TC + ABC

DETAILED DESCRIPTION:
In recent years mayor progress has been made in therapeutic approaches with the introduction of HAART, which has meant a huge fall in morbidity-mortality in Western countries.

However, despite having a variety of potent HAART combinations, some patients do not obtain adequate suppression. The causes of virological failure are complex, and one of the most significant factors is the incomplete compliance with the prescribed dosage of highly-active antiretroviral therapy (HAART). The development of fixed dose combination products is most commonly used to help simplify the dosages and improve treatment compliance.

One of the main problems associated with the treatment of HIV infection is the change in body structure, generally grouped under the term of lipodystrophy. These usually include fat accumulation in the stomach, or abdominal girth, and, even worse, atrophy in the face, arms, and legs. It is usually associated with metabolic disorders, with increased levels of triglycerides, cholesterol and/or insulin resistance.

The incidence of lipodystrophy increases progressively over time in patients starting treatment with antiretroviral agents. It is estimated that, after 2 years of treatment, 20%-30% of patients experience moderate or severe lipodystrophy.

Trizivir® is a combination of three antiretroviral agents: Abacavir, Lamivudine and Zidovudine in a tablet. All of them belong to the group of nucleoside/nucleotide analogue reverse transcriptase inhibitors (NRTIs.

The main advantage of Trizivir is the possibility of simplifying antiretroviral treatment. Multiple studies have been performed showing that simplification of HAART with Trizivir enhances compliance and improves quality of life in patients maintaining the efficacy of previous antiretroviral treatments.

Kaletra® (lopinavir+ritonavir) is a combination of two protease inhibitors: lopinavir plus a low dose of ritonavir, enhancing the action of the former.

Previous studies have shown that most patients treated with Kaletra monotherapy have an undetectable viral load after 48 weeks. Monotherapy failures were not associated with the development of primary resistance mutations.

To date the development of lipoatrophy appears to occur more frequently in patients with a NRTI- containing regimen. The combination of abacavir, zidovudine and lamivudine has been investigated in patients naive to antiretroviral treatments and in patients already treated with NRTIs.

In this setting, we designed this clinical trial to establish the potential benefit of Kaletra in monotherapy for the prevention of lipoatrophy. For this purpose, we will compare keeping on treatment with TZV in patients with viral suppression vs switching to Kaletra in monotherapy in order to prevent fat changes.

Since the purpose of the study is to establish the ability of Kaletra to prevent the development of and exclude patients with acute intolerance to Kaletra, the patients assigned to the experimental group will be treated for 4 weeks with Trizivir and Kaletra before switching to Kaletra monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV 1 documented by positive HIV 1 antibody test and/or positive PCR test confirmed for HIV 1 RNA.
* Patients on treatment with Trizivir with an undetectable viral burden defined as < 50 copies/ml in the past 6 months.
* Men or women aged ≥ 18 years.
* CD4 cell count ≥ 200 cells/μl.
* For women of child bearing age, a negative urine pregnancy test at the screening visit.
* Patients giving their written informed consent before completing any study specific screening procedure.

Exclusion Criteria:

* Patients with previously failed therapy with protease inhibitors (PI) or those receiving sub optimum therapy with nucleoside analogue reverse transcriptase inhibitors (NRTI) for the study disease.
* Presence of lipoatrophy defined by the investigator (any grade) or by the patient (in this case, at least two sites of mild degree or one of at least moderate degree).
* Known history of drug addiction or chronic use of alcohol that, in the investigator's opinion, contraindicates participation in the study.
* Pregnant or nursing women or women of child bearing age not using an adequate contraceptive method according to the investigator's criterion.
* Current active opportunistic infection or documented infection in the 4 weeks prior to screening.
* Renal disease with creatinine clearance < 50 ml/min.
* Concomitant use of nephrotoxic or immunosuppressive agents.
* Patient currently treated with systemic corticosteroids, interleukine 2, or chemotherapy.
* Patients treated with other investigational agents.
* Patients with acute hepatitis.
* Any disease that, at the criterion in the investigator, contraindicates the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Limb Fat changes measured by DEXA | 48 weeks

SECONDARY OUTCOMES:
20 % loss peripheral fat measured by DEXA | 96 weeks
Perception of change on body fat by physician and patient. | 96 weeks
Lipohypertrophy | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Iribarren, Study Chair — Hospital de Donostia
Locations (7):
- Spain (7):
  - Hospital Ntra.Sra. de Zumarraga, Zumarraga, Guipuzcua
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital de Donostia, Donostia / San Sebastian, San Sebastian
  - Hospital de Basurto, Bilbao, Vizcaya
  - H. Son Dureta, Mallorca